CLINICAL TRIAL: NCT00339924
Title: Physicians' Understanding of Human Genetic Variation
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905196; 05-HG-N196
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Genetics
Keywords: Clinical Decision-Making; Physician Bias; Genetics; Race; Ethnicity; Natural History; Human Genetic Variation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Currently practicing, board certified general internists, both allopathic and osteopathic, whose offices are in the United States.

SUMMARY:
This study will develop a survey instrument to measure primary care physicians' knowledge of the variation in human genetics, their beliefs about biologic and genetic differences according to patients' race and ethnicity, and how that knowledge is used in their clinical decision making.

Genomics research today is such that primary care physicians will be responsible for translating new genetic knowledge, drug therapies, and single and multiplex genetic testing into clinical practice.

Physicians who are board certified general internists, including those who practice and teach in research and teaching hospitals in urban areas of the United States, may be eligible for this study. Participants will be recruited through invitation and information letters mailed to leaders of local chapters of physician organizations, through letters and e-mail sent to qualifying general internists in databases, and through e-mail sent to academic physicians who practice or teach medicine at medical schools that meet the inclusion criteria. The number of participants is estimated at 96 in the first phase of the study. The researchers are especially interested in general internists who provide general and preventative health care services to patients of various racial, ethnic, and ancestral backgrounds. This study will use qualitative methods-focus groups and semistructured interviews-and quantitative methods. Two pilot focus group sessions, with about eight members each, are planned for Washington, D.C. Other settings for the study are Atlanta, Detroit, Los Angeles, and Philadelphia. Those locations were selected based on population density, availability of several teaching hospitals with diverse patient populations, availability of physicians meeting the study requirements, and the need to address important regions nationwide.

The focus groups will be separated by region and self-identified race-for example, one group consisting of African American internists from Atlanta and another of white internists from Atlanta. The facilitator will be a general internist of the same race. Each focus group session, to last about 90 minutes, will be audiotaped and transcribed verbatim. Data from the focus groups will be analyzed for themes and phrases, and a scale will be developed to assess responses. Then the scale will be reviewed by two panels of experts. One panel will be experts in genetics and human genetic variation, and the other will be social scientists and survey researchers who are experts in developing surveys. For the semistructured interviews, two physicians who participated in a given focus group will be invited to participate, based on their engagement in the discussion and interest in the project. This will be a face-to-face interview of 60 to 90 minutes. A total of 32 interviews will be conducted. After the scale is revised, a second pilot study will be done. For that study, 3,500 primary care physicians will be invited to participate in a web-based survey by using the scale. It is anticipated that there will be sufficient sample size to examine the properties of the scale. The proposed timetable for the study is 2 years.

Benefits from participating in the study include participants' increased understanding of human genetic variation and awareness of how other physicians understand and use race and ethnicity in their practice of medicine. Also, information gained will be useful to improve physicians' training. There will be compensation for participation. Each physician will receive $150, and those who participate in both the focus group and semistructured interview will receive $150 for each session.

...

DETAILED DESCRIPTION:
In recognition of the emerging social and scientific research related to assessing the complex relationships between self-identified race, ancestral origin and the genetic components of diseases, it is important to study physicians and other health professionals knowledge of human genetic variation and how they interpret and apply race, ethnicity and human genetic variation in their clinical decision making. Primary care physicians will be responsible for the translation of new genomic knowledge, including the use of pharmacogenomic and multiplex genetic testing in clinical practice. Understanding health professionals knowledge, beliefs and practices will provide important data for furthering health services and research. The Physicians Understanding of Human Genetic Variation study (PUHGV) is a three-phase, mixed-method study using both qualitative (focus groups and semi-structured interviews) and quantitative methods (web-based survey). The first phase of the study used qualitative methods to investigate racial and ethnic differences in how physicians understand and use genetics, race and ethnicity in their practice and to assist in developing the Health Professionals Genetic Education Needs Exploration survey instrument (HP GENE). Bonham and Sellers developed and piloted the Human Genetic Variation-Health Professionals Knowledge, Beliefs, and Use Scales (HGV-HP) to measure physicians knowledge of human genetic variation (HGV-HP Knowledge), beliefs about biologic and genetic differences based upon their patients race and ethnicity (HGV-HP Beliefs), and use of these constructs in their clinical decision making approaches (HGV-HP Use). The HGV-HP Scales are a component of the larger HP GENE survey instrument. The second phase of the study piloted these instruments with a random sample of United States general internists from diverse racial and ethnic backgrounds and geographic areas of the United States to assess the psychometric properties of the scales and investigate the role of incentives in recruiting physicians to participate in web surveys. Informed by the pilot testing of the instrument, the third phase of this study is to conduct a national survey using the instrument and scales with health professionals from different health disciplines.

ELIGIBILITY:
* INCLUSION CRITERIA:

The population of interest for this phase of the study are currently practicing, board certified general internists, both allopathic and osteopathic, whose offices are in the United States. Investigators have selected this population for multiple reasons. General internists are on the frontlines of health care delivery and have become increasingly more responsible for the translation of genomic knowledge into clinical practice.

Further, selecting general internists for this phase of the study is consistent with populations included in Phases I and II of the study. Lastly, limiting our pool of potential respondents to general internists helps to minimize costs associated with this study.

EXCLUSION CRITERIA:

We will exclude physicians with addresses outside of the continental United States, as well as, physicians who are not in active practice (see patients <10% of their time), deceased, or retired prior to randomly selecting the sample. Because questions surrounding clinical decision making are a key component of this survey, it is imperative that we only include practicing physicians in the sample.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest for this phase of the study are currently practicing, board certified general internists, both allopathic and osteopathic, whose offices are in the United States.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2005-07-11; Primary Completion 2012-04-13 (Actual); Study Completion 2012-04-13 (Actual)

PRIMARY OUTCOMES:
Knowledge and understanding | Ongoing
  The objective of this study is to investigate how health professionals understand and use genomics in clinical practice including their knowledge and understanding of human genetic variation, race, and ethnicity in disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Vence L Bonham, J.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Collins FS, Green ED, Guttmacher AE, Guyer MS; US National Human Genome Research Institute. A vision for the future of genomics research. Nature. 2003 Apr 24;422(6934):835-47. doi: 10.1038/nature01626. Epub 2003 Apr 14. No abstract available. PMID 12695777
- [Background] Grumbach K, Bodenheimer T. A primary care home for Americans: putting the house in order. JAMA. 2002 Aug 21;288(7):889-93. doi: 10.1001/jama.288.7.889. PMID 12186609
- [Background] Schwartz RS. Racial profiling in medical research. N Engl J Med. 2001 May 3;344(18):1392-3. doi: 10.1056/NEJM200105033441810. No abstract available. PMID 11333999